CLINICAL TRIAL: NCT02637557
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-range-finding Trial of IW-3718 Administered Orally for 8 Weeks to Patients With Symptomatic Gastroesophageal Reflux Disease Not Completely Responsive to Proton Pump Inhibitors
Brief Title: A Trial of IW-3718 for 8 Weeks in Patients With Symptomatic Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICP-3718-202
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Placebo Comparator): Matching placebo twice daily
  Interventions: Drug: Matching Placebo; Drug: PPI
- 500 mg IW-3718 (Experimental): 500 mg IW-3718 twice daily
  Interventions: Drug: IW-3718; Drug: PPI
- 1000 mg IW-3718 (Experimental): 1000 mg IW-3718 twice daily
  Interventions: Drug: IW-3718; Drug: PPI
- 1500 mg IW-3718 (Experimental): 1500 mg IW-3718 twice daily
  Interventions: Drug: IW-3718; Drug: PPI

INTERVENTIONS:
Drug: IW-3718
  Arms: 1000 mg IW-3718; 1500 mg IW-3718; 500 mg IW-3718
Drug: Matching Placebo
  Arms: Control
Drug: PPI — All participants were taking a standard dose QD PPI (dexlansoprazole, esomeprazole, esomeprazole magnesium, lansoprazole, omeprazole, pantoprazole, pantoprazole sodium sesquihydrate, rabeprazole or rabeprazole sodium) during the study.

SUMMARY:
The objectives of this study are to evaluate the safety, efficacy, and dose-response relationship of IW-3718 administered orally to participants who have GERD and continue to experience GERD symptoms while receiving once-daily (QD), standard-dose proton pump inhibitors (PPIs).

ELIGIBILITY:
Inclusion Criteria:

* Patient is an ambulatory, community-dwelling male or nonpregnant female and is at least 18 years old at the Screening Visit. Lactating females must agree not to breastfeed.
* Patient has a diagnosis of GERD and reports experiencing GERD symptoms (heartburn or regurgitation) on ≥ 4 days per week during the 8 weeks before the Screening Visit while taking standard QD PPI therapy.

Exclusion Criteria:

* Patient may not meet any of the excluded conditions specified in the protocol
* Patient has any alarm symptoms including but not limited to GI bleeding, anemia, vomiting, dysphagia, or unexpected weight loss any time during the Screening or Pretreatment Periods
* Patient has a history of clinically significant hypersensitivity or allergies to any of the excipients contained in the study medication (active or placebo).

NOTE: Additional inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Lane, Study Director — Ironwood Pharmaceuticals, Inc.
Locations (57):
- United States (57):
  - IW-3718 Investigator, Dothan, Alabama
  - IW-3718 Investigator, Phoenix, Arizona
  - IW-3718 Investigator, Tucson, Arizona
  - IW-3718 Investigator, North Little Rock, Arkansas
  - IW-3718 Investigator, Anaheim, California
  - IW-3718 Investigator, Carmichael, California
  - IW-3718 Investigator, Chula Vista, California
  - IW-3718 Investigator, La Mirada, California
  - IW-3718 Investigator, Mission Hills, California
  - IW-3718 Investigator, Newport Beach, California
  - IW-3718 Investigator, Oakland, California
  - IW-3718 Investigator, Sacramento, California
  - IW-3718 Investigator, San Diego, California
  - IW-3718 Investigator, Bristol, Connecticut
  - IW-3718 Investigator, Waterbury, Connecticut
  - IW-3718 Investigator, DeLand, Florida
  - IW-3718 Investigator, Hollywood, Florida
  - IW-3718 Investigator, Inverness, Florida
  - IW-3718 Investigator, Jupiter, Florida
  - IW-3718 Investigator, Lauderdale Lakes, Florida
  - IW-3718 Investigator, Miami, Florida
  - IW-3718 Investigator, Miami Lakes, Florida
  - IW-3718 Investigator, Port Orange, Florida
  - IW-3718 Investigator, Clive, Iowa
  - IW-3718 Investigator, Bowling Green, Kentucky
  - IW-3718 Investigator, Monroe, Louisiana
  - IW-3718 Investigator, Annapolis, Maryland
  - IW-3718 Investigator, Baltimore, Maryland
  - IW-3718 Investigator, Chevy Chase, Maryland
  - IW-3718 Investigator, Chesterfield, Michigan
  - IW-3718 Investigator, Wyoming, Michigan
  - IW-3718 Investigator, Las Vegas, Nevada
  - IW-3718 Investigator, Reno, Nevada
  - IW-3718 Investigator, Egg Harbor, New Jersey
  - IW-3718 Investigator, Great Neck, New York
  - IW-3718 Investigator, Kew Gardens, New York
  - IW-3718 Investigator, New York, New York
  - IW-3718 Investigator, Asheville, North Carolina
  - IW-3718 Investigator, Raleigh, North Carolina
  - IW-3718 Investigator, Fargo, North Dakota
  - IW-3718 Investigator, Cleveland, Ohio
  - IW-3718 Investigator, Columbus, Ohio
  - IW-3718 Investigator, Lima, Ohio
  - IW-3718 Investigator, Norman, Oklahoma
  - IW-3718 Investigator, Oklahoma City, Oklahoma
  - IW-3718 Investigator, Pittsburgh, Pennsylvania
  - IW-3718 Investigator, Charleston, South Carolina
  - IW-3718 Investigator, Chattanooga, Tennessee
  - IW-3718 Investigator, Germantown, Tennessee
  - IW-3718 Investigator, Nashville, Tennessee
  - IW-3718 Investigator, El Paso, Texas
  - IW-3718 Investigator, Houston, Texas
  - IW-3718 Investigator, San Antonio, Texas
  - IW-3718 Investigator, Sandy City, Utah
  - IW-3718 Investigator, South Ogden, Utah
  - IW-3718 Investigator, Christiansburg, Virginia
  - IW-3718 Investigator, Lynchburg, Virginia

REFERENCES:
- [Derived] Vaezi MF, Fass R, Vakil N, Reasner DS, Mittleman RS, Hall M, Shao JZ, Chen Y, Lane L, Gates AM, Currie MG. IW-3718 Reduces Heartburn Severity in Patients With Refractory Gastroesophageal Reflux Disease in a Randomized Trial. Gastroenterology. 2020 Jun;158(8):2093-2103. doi: 10.1053/j.gastro.2020.02.031. Epub 2020 Feb 22. PMID 32092310
- [Derived] Andrae DA, Hanlon J, Cala ML, Scippa K, Graham C, Witherspoon B, Shao JZ, Reasner D. Evaluation and Validation of the Modified Reflux Symptom Questionnaire-Electronic Diary in Patients With Persistent Gastroesophageal Reflux Disease. Clin Transl Gastroenterol. 2020 Jan;11(1):e00117. doi: 10.14309/ctg.0000000000000117. PMID 31977454

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo BID: Matching placebo twice daily (BID)
- 500 mg IW-3718 BID: 500 mg IW-3718 BID
- 1000 mg IW-3718 BID: 1000 mg IW-3718 BID
- 1500 mg IW-3718 BID: 1500 mg IW-3718 BID
Period: Overall Study
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Started | 71 | 71 | 71 | 69
Completed | 63 | 66 | 62 | 62
Not Completed | 8 | 5 | 9 | 7
Not completed — Adverse Event | 3 | 1 | 3 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Population: modified Intent-to-Treat Population: all randomized participants who received at least one dose of study treatment.
Groups:
- Placebo BID: Matching placebo BID
- Total: Total of all reporting groups
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID | Total
Number analyzed (Participants) | 70 | 71 | 71 | 68 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (12.9) | 51.4 (13.3) | 50.1 (11.2) | 49.4 (12.3) | 50.1 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 46 | 43 | 39 | 171
  Male | 27 | 25 | 28 | 29 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 23 | 15 | 17 | 64
  Not Hispanic or Latino | 61 | 48 | 56 | 51 | 216
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 0 | 1 | 3
  Black or African American | 12 | 8 | 9 | 10 | 39
  Caucasian | 54 | 62 | 62 | 54 | 232
  Other, Not Specified | 2 | 1 | 0 | 3 | 6
Weekly Heartburn Severity Score (WHSS) [Mean (Standard Deviation); unit: score on a scale] — The WHSS for an analysis week was defined as the average of available Daily Heartburn Severity Scale (DHSS) during that week. DHSS was defined as the maximum on a 6-point scale (0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe) of the 3 items measuring heartburn ("Heartburn," "Burning feeling behind breastbone or in the center of the upper stomach," and "Pain behind breastbone or in the center of the upper stomach") from a particular day.
  Baseline was derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization.
  score on a scale | 3.18 (0.64) | 3.19 (0.72) | 3.12 (0.64) | 3.19 (0.71) | 3.17 (0.68)
Modified Reflux Symptom Questionnaire - Electronic Diary (mRESQ-eD) Item 'Heartburn Severity' [Mean (Standard Deviation); unit: units on a scale] — The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the severity of their heartburn over the past 24 hours on a 6-point scale: 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe.
  Baseline was derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization.
  units on a scale | 3.08 (0.63) | 3.01 (0.66) | 3.00 (0.64) | 3.08 (0.66) | 3.04 (0.65)
mRESQ-eD Item 'Burning Feeling Behind Breastbone or Center of Upper Stomach Severity' [Mean (Standard Deviation); unit: units on a scale] — The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the severity of their burning feeling behind the breastbone or in the center of the upper stomach over the past 24 hours on a 6-point scale: 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe.
  Baseline was derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization.
  units on a scale | 2.85 (0.82) | 2.91 (0.82) | 2.77 (0.82) | 2.98 (0.78) | 2.88 (0.81)
mRESQ-eD Item 'Pain Behind Breastbone or Center of Upper Stomach Severity' [Mean (Standard Deviation); unit: units on a scale] — The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the severity of their pain behind the breastbone or in the center of the upper stomach over the past 24 hours on a 6-point scale: 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe.
  Baseline was derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization.
  units on a scale | 2.73 (0.87) | 2.80 (0.89) | 2.57 (0.95) | 2.85 (0.91) | 2.74 (0.91)
mRESQ-eD Item 'Difficulty Swallowing Severity' [Mean (Standard Deviation); unit: units on a scale] — The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the severity of their difficulty swallowing over the past 24 hours on a 6-point scale: 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe.
  Baseline was derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization.
  units on a scale | 1.71 (1.19) | 1.81 (1.27) | 2.15 (1.27) | 2.05 (1.17) | 1.93 (1.23)
mRESQ-eD Item 'Hoarseness Severity' [Mean (Standard Deviation); unit: units on a scale] — The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the severity of their hoarseness over the past 24 hours on a 6-point scale: 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe.
  Baseline was derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization.
  units on a scale | 1.75 (1.18) | 1.81 (1.31) | 2.00 (1.35) | 1.81 (1.31) | 1.84 (1.29)
mRESQ-eD Item 'Cough Severity' [Mean (Standard Deviation); unit: units on a scale] — The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the severity of their cough over the past 24 hours on a 6-point scale: 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe.
  Baseline was derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization.
  units on a scale | 1.78 (1.27) | 2.11 (1.26) | 2.21 (1.23) | 2.16 (1.22) | 2.07 (1.25)
mRESQ-eD Item 'Regurgitation Frequency' [Mean (Standard Deviation); unit: units on a scale] — The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the frequency of their regurgitation (liquid or food moving upwards towards the throat or mouth) over the past 24 hours on a 5-point scale: 0=Never, 1= Rarely, 2=Sometimes, 3=Often, 4=Very often.
  Baseline was derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization.
  units on a scale | 2.03 (0.99) | 2.29 (0.80) | 2.11 (0.97) | 2.19 (0.88) | 2.15 (0.92)
mRESQ-eD Item 'Acid or Bitter Taste Frequency' [Mean (Standard Deviation); unit: units on a scale] — The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the frequency of an acid or bitter taste in the mouth over the past 24 hours on a 5-point scale: 0=Never, 1= Rarely, 2=Sometimes, 3=Often, 4=Very often.
  Baseline was derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization.
  units on a scale | 2.09 (1.06) | 2.25 (0.88) | 2.21 (0.98) | 2.19 (1.01) | 2.18 (0.98)
mRESQ-eD Item 'Coughing Frequency' [Mean (Standard Deviation); unit: units on a scale] — The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the frequency of their cough over the past 24 hours on a 5-point scale: 0=Never, 1= Rarely, 2=Sometimes, 3=Often, 4=Very often.
  Baseline was derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization.
  units on a scale | 1.65 (1.10) | 1.91 (1.06) | 1.96 (0.99) | 1.96 (1.00) | 1.87 (1.04)
mRESQ-eD Item 'Burping Frequency' [Mean (Standard Deviation); unit: units on a scale] — The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the frequency of their burping over the past 24 hours on a 5-point scale: 0=Never, 1= Rarely, 2=Sometimes, 3=Often, 4=Very often.
  Baseline was derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization.
  units on a scale | 2.26 (1.04) | 2.21 (0.91) | 2.33 (0.85) | 2.51 (0.90) | 2.33 (0.93)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 8 in Weekly Heartburn Severity Score (WHSS)
Description: The WHSS for an analysis week was defined as the average of available DHSS during that week. DHSS was defined as the maximum on a 6-point scale (0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe) of the 3 items measuring heartburn ( "Heartburn," "Burning feeling behind breastbone or in the center of the upper stomach," and "Pain behind breastbone or in the center of the upper stomach,") from a particular day. A negative change from Baseline indicates improvement.
Time Frame: Baseline (derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization), Week 8
Population: modified Intent-to-Treat Population: all randomized participants who received at least one dose of study treatment with values both at baseline and during the Treatment Period.
Measure: Least Squares Mean (Standard Error); unit: percentage change in score
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
percentage change in score | -46.026 (4.078) | -48.978 (4.019) | -55.063 (4.024) | -57.969 (4.108)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Test type: Superiority; p = 0.6065, ANCOVA — P-value based on a pairwise comparison versus placebo in an ANCOVA model with fixed effect terms for treatment group and esophagitis stratum and baseline value as covariate; LS Mean Difference = -2.952, 95% CI 2-sided [-14.222 to 8.318]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Test type: Superiority; p = 0.1160, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -9.036, 95% CI 2-sided [-20.318 to 2.245]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.0400, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -11.943, 95% CI 2-sided [-23.334 to -0.551]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID vs 1000 mg IW-3718 BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.0225, trend test — Dose trend test performed using linear contrast statement

2. Secondary Outcome: Percent Change From Baseline to Week 4 in WHSS
Description: as for outcome 1
Time Frame: Baseline (derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization), Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage change in score
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
percentage change in score | -38.883 (3.733) | -42.594 (3.679) | -41.622 (3.683) | -47.486 (3.761)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Test type: Superiority; p = 0.4795, ANCOVA — P-values are based on a pairwise comparison versus placebo in an ANCOVA model with fixed effect terms for treatment group and esophagitis stratum and baseline value as covariate; LS Mean Difference = -3.711, 95% CI 2-sided [-14.028 to 6.606]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Test type: Superiority; p = 0.6020, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -2.739, 95% CI 2-sided [-13.066 to 7.588]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.1055, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -8.602, 95% CI 2-sided [-19.030 to 1.826]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID vs 1000 mg IW-3718 BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.1387, trend test — Dose trend test performed using linear contrast statement

3. Secondary Outcome: Change From Baseline to Week 8 in WHSS
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
score on a scale | -1.459 (0.129) | -1.517 (0.127) | -1.713 (0.127) | -1.876 (0.130)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Test type: Superiority; p = 0.7488, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.058, 95% CI 2-sided [-0.415 to 0.299]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Test type: Superiority; p = 0.1627, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.254, 95% CI 2-sided [-0.611 to 0.103]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.0237, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.417, 95% CI 2-sided [-0.777 to -0.056]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID vs 1000 mg IW-3718 BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.0130, trend test — Dose trend test performed using linear contrast statement

4. Secondary Outcome: Change From Baseline to Week 4 in WHSS
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
score on a scale | -1.261 (0.115) | -1.313 (0.113) | -1.308 (0.113) | -1.517 (0.115)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Test type: Superiority; p = 0.7470, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.052, 95% CI 2-sided [-0.369 to 0.265]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Test type: Superiority; p = 0.7699, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.047, 95% CI 2-sided [-0.364 to 0.270]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.1157, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.257, 95% CI 2-sided [-0.577 to 0.064]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID vs 1000 mg IW-3718 BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.1374, trend test — Dose trend test performed using linear contrast statement

5. Secondary Outcome: Percentage of Participants Who Are Overall Heartburn Responders
Description: An overall heartburn responder is a participant who is a weekly heartburn responder for at least 4 of the 8 treatment weeks and for at least 1 of the final 2 treatment weeks (i.e., Week 7 and Week 8). A weekly heartburn responder is a participant with a decrease of >= 30% from baseline in WHSS (see Outcome Measure 1 for description of WHSS). A participant who reported heartburn severity for less than 4 days during a week was not considered a responder for that week.
Time Frame: Week 8
Population: modified Intent-to-Treat Population: all randomized participants who received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 70 | 71 | 71 | 68
percentage of participants | 54.3 [41.9 to 66.3] | 52.1 [39.9 to 64.1] | 62.0 [49.7 to 73.2] | 66.2 [53.7 to 77.2]
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Test type: Superiority; p = 0.7903, Cochran-Mantel-Haenszel — Odds ratio, 95% confidence interval (CI) for the odds ratio and p-value vs. placebo are obtained from the Cochran-Mantel-Haenszel (CMH) tests controlling for esophagitis status; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.47 to 1.77]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Test type: Superiority; p = 0.3518, Cochran-Mantel-Haenszel — Odds ratio, 95% CI for the odds ratio and p-value vs. placebo are obtained from the CMH tests controlling for esophagitis status; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.70 to 2.71]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.1544, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.83 to 3.26]

6. Secondary Outcome: Percentage of Participants With a DHSS of No More Than Very Mild (≤ 1) on Any Day During Week 8
Description: DHSS was defined as the maximum on a 6-point scale (0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe) of the 3 items measuring heartburn ( "Heartburn," "Burning feeling behind breastbone or in the center of the upper stomach," and "Pain behind breastbone or in the center of the upper stomach,") from a particular day. A participant who reported heartburn severity for less than 4 days during a week was not considered a responder for that week.
Time Frame: Week 8
Population: modified Intent-to-Treat Population: all randomized participants who received at least one dose of study treatment with values both at baseline and given treatment week.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 70 | 71 | 71 | 68
percentage of participants | 28.6 [18.4 to 40.6] | 18.3 [10.1 to 29.3] | 29.6 [19.3 to 41.6] | 38.2 [26.7 to 50.8]
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Test type: Superiority; p = 0.1489, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.25 to 1.23]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Test type: Superiority; p = 0.8891, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.51 to 2.19]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.2237, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 2]; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.76 to 3.20]

7. Secondary Outcome: Percentage of Participants With a DHSS of No More Than Very Mild (≤ 1) on Any Day During Week 4
Description: as for outcome 6
Time Frame: Week 4
Population: modified Intent-to-Treat Population: all randomized participants who received at least one dose of study treatment with values at both baseline and given treatment week.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 70 | 71 | 71 | 68
percentage of participants | 12.9 [6.1 to 23.0] | 15.5 [8.0 to 26.0] | 22.5 [13.5 to 34.0] | 22.1 [12.9 to 33.8]
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Test type: Superiority; p = 0.6566, Cochran-Mantel-Haenszel — Odds ratio, 95% CI (Confidence Interval) for the Odds Ratio and p-value vs. placebo are obtained from the CMH tests controlling for esophagitis status; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.48 to 3.18]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Test type: Superiority; p = 0.1280, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 2.01, 95% CI 2-sided [0.81 to 4.98]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.1463, Cochran-Mantel-Haenszel — [p-value comment as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.97, 95% CI 2-sided [0.79 to 4.91]

8. Secondary Outcome: Change From Baseline in the Number of Days Where DHSS Was No More Than Very Mild (≤ 1) During Week 8
Description: DHSS was defined as the maximum on a 6-point scale (0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe) of the 3 items measuring heartburn ( "Heartburn," "Burning feeling behind breastbone or in the center of the upper stomach," and "Pain behind breastbone or in the center of the upper stomach,") from a particular day.
Time Frame: Week 8
Population: modified Intent-to-Treat Population: all randomized participants who received at least one dose of study treatment with values at both baseline and treatment week.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 62 | 66 | 63 | 62
days | 2.998 (0.358) | 2.700 (0.347) | 3.250 (0.355) | 3.510 (0.359)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Test type: Superiority; p = 0.5504, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.298, 95% CI 2-sided [-1.279 to 0.683]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Test type: Superiority; p = 0.6177, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.252, 95% CI 2-sided [-0.741 to 1.244]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.3138, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.513, 95% CI 2-sided [-0.488 to 1.513]

9. Secondary Outcome: Change From Baseline in the Number of Days Where DHSS Was No More Than Very Mild (≤ 1) During Week 4
Description: as for outcome 8
Time Frame: Week 4
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 64 | 70 | 67 | 68
days | 2.275 (0.336) | 2.294 (0.322) | 2.694 (0.329) | 2.736 (0.327)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Test type: Superiority; p = 0.9675, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.019, 95% CI 2-sided [-0.897 to 0.935]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Test type: Superiority; p = 0.3741, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.419, 95% CI 2-sided [-0.507 to 1.345]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.3275, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.461, 95% CI 2-sided [-0.464 to 1.385]

10. Secondary Outcome: Change From Baseline Over Time in the Weekly Average of Modified Reflux Symptom Questionnaire - Electronic Diary (mRESQ-eD) Item 'Heartburn Severity'
Description: The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the severity of their heartburn over the past 24 hours on a 6-point scale: 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe. Daily scores were averaged each week. A negative change from Baseline indicates improvement.
Time Frame: Baseline (derived from the eDiary daily data collected from 7 days before randomization up to the time of randomization), Weeks 1, 2, 3, 4, 5, 6, 7, 8
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
units on a scale
  Week 1 | -0.655 (0.090) | -0.632 (0.089) | -0.531 (0.089) | -0.673 (0.091)
  Week 2 | -0.994 (0.102) | -0.974 (0.101) | -0.977 (0.101) | -1.102 (0.103)
  Week 3 | -1.092 (0.109) | -1.141 (0.107) | -1.153 (0.107) | -1.350 (0.109)
  Week 4 | -1.263 (0.112) | -1.281 (0.110) | -1.259 (0.110) | -1.498 (0.112)
  Week 5 | -1.284 (0.120) | -1.301 (0.119) | -1.339 (0.119) | -1.677 (0.121)
  Week 6 | -1.396 (0.121) | -1.343 (0.119) | -1.467 (0.119) | -1.744 (0.122)
  Week 7 | -1.392 (0.127) | -1.350 (0.125) | -1.436 (0.125) | -1.693 (0.128)
  Week 8 | -1.404 (0.127) | -1.482 (0.126) | -1.666 (0.126) | -1.807 (0.128)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.8560, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.023, 95% CI 2-sided [-0.226 to 0.272]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.3301, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.124, 95% CI 2-sided [-0.126 to 0.373]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.8845, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.019, 95% CI 2-sided [-0.270 to 0.233]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.8879, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.020, 95% CI 2-sided [-0.262 to 0.303]
Statistical Analysis 5: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.9072, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.017, 95% CI 2-sided [-0.266 to 0.299]
Statistical Analysis 6: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.4573, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.108, 95% CI 2-sided [-0.393 to 0.177]
Statistical Analysis 7: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.7476, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.049, 95% CI 2-sided [-0.350 to 0.251]
Statistical Analysis 8: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.6873, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.062, 95% CI 2-sided [-0.362 to 0.239]
Statistical Analysis 9: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.0952, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.258, 95% CI 2-sided [-0.562 to 0.045]
Statistical Analysis 10: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.9111, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.018, 95% CI 2-sided [-0.326 to 0.291]
Statistical Analysis 11: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.9772, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.004, 95% CI 2-sided [-0.304 to 0.313]
Statistical Analysis 12: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.1390, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.235, 95% CI 2-sided [-0.546 to 0.077]
Statistical Analysis 13: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.9215, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.017, 95% CI 2-sided [-0.349 to 0.316]
Statistical Analysis 14: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.7453, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.055, 95% CI 2-sided [-0.388 to 0.278]
Statistical Analysis 15: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.0220, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.393, 95% CI 2-sided [-0.729 to -0.057]
Statistical Analysis 16: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.7561, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.053, 95% CI 2-sided [-0.282 to 0.387]
Statistical Analysis 17: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.6758, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.071, 95% CI 2-sided [-0.406 to 0.263]
Statistical Analysis 18: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.0434, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.348, 95% CI 2-sided [-0.686 to -0.010]
Statistical Analysis 19: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.8123, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.042, 95% CI 2-sided [-0.308 to 0.392]
Statistical Analysis 20: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.8038, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.044, 95% CI 2-sided [-0.394 to 0.306]
Statistical Analysis 21: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.0954, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.300, 95% CI 2-sided [-0.654 to 0.053]
Statistical Analysis 22: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.6649, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.078, 95% CI 2-sided [-0.430 to 0.275]
Statistical Analysis 23: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.1448, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.262, 95% CI 2-sided [-0.614 to 0.091]
Statistical Analysis 24: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.0264, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.403, 95% CI 2-sided [-0.759 to -0.048]

11. Secondary Outcome: Change From Baseline Over Time in the Weekly Average of mRESQ-eD Item 'Burning Feeling Behind Breastbone or Center of Upper Stomach Severity'
Description: The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the severity of their burning feeling behind the breastbone or in the center of the upper stomach over the past 24 hours on a 6-point scale: 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe. Daily scores were averaged each week. A negative change from baseline indicates improvement.
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
units on a scale
  Week 1 | -0.638 (0.089) | -0.536 (0.087) | -0.492 (0.088) | -0.675 (0.089)
  Week 2 | -0.998 (0.103) | -0.918 (0.101) | -0.970 (0.102) | -1.116 (0.104)
  Week 3 | -1.040 (0.108) | -1.074 (0.106) | -1.112 (0.107) | -1.385 (0.109)
  Week 4 | -1.199 (0.113) | -1.246 (0.112) | -1.316 (0.112) | -1.497 (0.114)
  Week 5 | -1.226 (0.120) | -1.287 (0.118) | -1.323 (0.118) | -1.648 (0.121)
  Week 6 | -1.357 (0.119) | -1.297 (0.117) | -1.450 (0.117) | -1.733 (0.120)
  Week 7 | -1.310 (0.124) | -1.359 (0.122) | -1.424 (0.122) | -1.676 (0.125)
  Week 8 | -1.329 (0.122) | -1.422 (0.120) | -1.627 (0.121) | -1.781 (0.123)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.4137, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.102, 95% CI 2-sided [-0.143 to 0.347]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.2395, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.147, 95% CI 2-sided [-0.098 to 0.392]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.7729, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.036, 95% CI 2-sided [-0.284 to 0.212]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.5824, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.079, 95% CI 2-sided [-0.205 to 0.363]
Statistical Analysis 5: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.8466, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.028, 95% CI 2-sided [-0.256 to 0.312]
Statistical Analysis 6: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.4192, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.118, 95% CI 2-sided [-0.405 to 0.169]
Statistical Analysis 7: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.8192, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.035, 95% CI 2-sided [-0.333 to 0.264]
Statistical Analysis 8: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.6320, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.073, 95% CI 2-sided [-0.372 to 0.226]
Statistical Analysis 9: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.0254, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.345, 95% CI 2-sided [-0.647 to -0.043]
Statistical Analysis 10: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.7689, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.047, 95% CI 2-sided [-0.360 to 0.266]
Statistical Analysis 11: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.4631, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.117, 95% CI 2-sided [-0.430 to 0.196]
Statistical Analysis 12: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.0651, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.298, 95% CI 2-sided [-0.615 to 0.019]
Statistical Analysis 13: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.7197, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.060, 95% CI 2-sided [-0.392 to 0.271]
Statistical Analysis 14: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.5649, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.097, 95% CI 2-sided [-0.428 to 0.234]
Statistical Analysis 15: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.0138, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.422, 95% CI 2-sided [-0.757 to -0.087]
Statistical Analysis 16: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.7202, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.060, 95% CI 2-sided [-0.269 to 0.388]
Statistical Analysis 17: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.5784, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.093, 95% CI 2-sided [-0.421 to 0.236]
Statistical Analysis 18: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.0266, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.376, 95% CI 2-sided [-0.708 to -0.044]
Statistical Analysis 19: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.7770, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.049, 95% CI 2-sided [-0.391 to 0.293]
Statistical Analysis 20: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.5121, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.114, 95% CI 2-sided [-0.456 to 0.228]
Statistical Analysis 21: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.0384, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.366, 95% CI 2-sided [-0.711 to -0.020]
Statistical Analysis 22: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.5876, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.093, 95% CI 2-sided [-0.431 to 0.245]
Statistical Analysis 23: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.0842, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.298, 95% CI 2-sided [-0.636 to 0.040]
Statistical Analysis 24: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.0098, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.452, 95% CI 2-sided [-0.793 to -0.110]

12. Secondary Outcome: Change From Baseline Over Time in the mRESQ-eD Item 'Pain Behind Breastbone or Center of Upper Stomach Severity'
Description: The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the severity of their pain behind the breastbone or in the center of the upper stomach over the past 24 hours on a 6-point scale: 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe. Daily scores were averaged each week. A negative change from baseline indicates improvement.
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
units on a scale
  Week 1 | -0.602 (0.089) | -0.548 (0.088) | -0.454 (0.089) | -0.626 (0.090)
  Week 2 | -0.921 (0.103) | -0.869 (0.101) | -0.934 (0.102) | -1.083 (0.103)
  Week 3 | -1.002 (0.110) | -1.008 (0.108) | -1.126 (0.109) | -1.313 (0.111)
  Week 4 | -1.185 (0.113) | -1.210 (0.111) | -1.244 (0.112) | -1.439 (0.114)
  Week 5 | -1.279 (0.119) | -1.230 (0.117) | -1.299 (0.118) | -1.578 (0.120)
  Week 6 | -1.343 (0.118) | -1.257 (0.117) | -1.367 (0.117) | -1.665 (0.119)
  Week 7 | -1.252 (0.122) | -1.303 (0.121) | -1.302 (0.121) | -1.638 (0.124)
  Week 8 | -1.289 (0.121) | -1.333 (0.119) | -1.525 (0.119) | -1.674 (0.122)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.6663, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.054, 95% CI 2-sided [-0.193 to 0.301]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.2400, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.148, 95% CI 2-sided [-0.100 to 0.396]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.8560, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.023, 95% CI 2-sided [-0.273 to 0.227]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.7209, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.051, 95% CI 2-sided [-0.232 to 0.335]
Statistical Analysis 5: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.9283, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.013, 95% CI 2-sided [-0.297 to 0.271]
Statistical Analysis 6: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.2659, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.162, 95% CI 2-sided [-0.449 to 0.124]
Statistical Analysis 7: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.9680, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.006, 95% CI 2-sided [-0.310 to 0.298]
Statistical Analysis 8: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.4213, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.125, 95% CI 2-sided [-0.429 to 0.180]
Statistical Analysis 9: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.0471, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.311, 95% CI 2-sided [-0.618 to -0.004]
Statistical Analysis 10: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.8769, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.025, 95% CI 2-sided [-0.337 to 0.288]
Statistical Analysis 11: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.7109, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.059, 95% CI 2-sided [-0.372 to 0.254]
Statistical Analysis 12: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.1146, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.254, 95% CI 2-sided [-0.570 to 0.062]
Statistical Analysis 13: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.7736, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.048, 95% CI 2-sided [-0.281 to 0.378]
Statistical Analysis 14: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.9059, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.020, 95% CI 2-sided [-0.350 to 0.310]
Statistical Analysis 15: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.0779, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.299, 95% CI 2-sided [-0.633 to 0.034]
Statistical Analysis 16: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.6068, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.086, 95% CI 2-sided [-0.241 to 0.412]
Statistical Analysis 17: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.8838, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.024, 95% CI 2-sided [-0.352 to 0.303]
Statistical Analysis 18: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.0556, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.323, 95% CI 2-sided [-0.653 to 0.008]
Statistical Analysis 19: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.7673, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.051, 95% CI 2-sided [-0.389 to 0.287]
Statistical Analysis 20: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.7709, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.050, 95% CI 2-sided [-0.389 to 0.289]
Statistical Analysis 21: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.0273, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.386, 95% CI 2-sided [-0.728 to -0.043]
Statistical Analysis 22: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.7950, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.044, 95% CI 2-sided [-0.378 to 0.289]
Statistical Analysis 23: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.1656, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.236, 95% CI 2-sided [-0.570 to 0.098]
Statistical Analysis 24: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.0254, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.385, 95% CI 2-sided [-0.722 to -0.048]

13. Secondary Outcome: Change From Baseline Over Time in the mRESQ-eD Item 'Difficulty Swallowing Severity'
Description: The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the severity of their difficulty swallowing over the past 24 hours on a 6-point scale: 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe. Daily scores were averaged each week. A negative change from baseline indicates improvement.
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
units on a scale
  Week 1 | -0.498 (0.075) | -0.405 (0.074) | -0.309 (0.074) | -0.519 (0.076)
  Week 2 | -0.618 (0.088) | -0.566 (0.086) | -0.611 (0.087) | -0.714 (0.088)
  Week 3 | -0.671 (0.094) | -0.675 (0.092) | -0.817 (0.092) | -1.022 (0.094)
  Week 4 | -0.737 (0.098) | -0.763 (0.096) | -0.810 (0.096) | -1.061 (0.098)
  Week 5 | -0.824 (0.098) | -0.850 (0.096) | -0.846 (0.096) | -1.156 (0.098)
  Week 6 | -0.883 (0.102) | -0.805 (0.100) | -0.961 (0.100) | -1.174 (0.102)
  Week 7 | -0.849 (0.107) | -0.756 (0.105) | -0.906 (0.106) | -1.166 (0.108)
  Week 8 | -0.864 (0.107) | -0.822 (0.105) | -0.989 (0.105) | -1.197 (0.107)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.3788, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.093, 95% CI 2-sided [-0.114 to 0.300]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.0761, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.189, 95% CI 2-sided [-0.020 to 0.397]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.8415, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.021, 95% CI 2-sided [-0.232 to 0.189]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.6719, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.052, 95% CI 2-sided [-0.190 to 0.294]
Statistical Analysis 5: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.9549, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.007, 95% CI 2-sided [-0.237 to 0.251]
Statistical Analysis 6: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.4408, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.096, 95% CI 2-sided [-0.342 to 0.149]
Statistical Analysis 7: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.9736, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.004, 95% CI 2-sided [-0.262 to 0.253]
Statistical Analysis 8: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.2703, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.146, 95% CI 2-sided [-0.405 to 0.114]
Statistical Analysis 9: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.0087, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.351, 95% CI 2-sided [-0.612 to -0.089]
Statistical Analysis 10: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.8480, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.026, 95% CI 2-sided [-0.295 to 0.243]
Statistical Analysis 11: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.5966, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.073, 95% CI 2-sided [-0.344 to 0.198]
Statistical Analysis 12: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.0203, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.324, 95% CI 2-sided [-0.596 to -0.051]
Statistical Analysis 13: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.8540, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.025, 95% CI 2-sided [-0.294 to 0.244]
Statistical Analysis 14: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.8757, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.022, 95% CI 2-sided [-0.293 to 0.250]
Statistical Analysis 15: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.0174, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.332, 95% CI 2-sided [-0.605 to -0.059]
Statistical Analysis 16: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.5831, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.078, 95% CI 2-sided [-0.202 to 0.358]
Statistical Analysis 17: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.5859, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.078, 95% CI 2-sided [-0.360 to 0.204]
Statistical Analysis 18: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.0447, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.291, 95% CI 2-sided [-0.575 to -0.007]
Statistical Analysis 19: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.5365, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.093, 95% CI 2-sided [-0.203 to 0.388]
Statistical Analysis 20: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.7067, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.057, 95% CI 2-sided [-0.355 to 0.241]
Statistical Analysis 21: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.0386, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.317, 95% CI 2-sided [-0.616 to -0.017]
Statistical Analysis 22: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.7804, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.042, 95% CI 2-sided [-0.253 to 0.336]
Statistical Analysis 23: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.4064, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.125, 95% CI 2-sided [-0.422 to 0.171]
Statistical Analysis 24: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.0289, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.333, 95% CI 2-sided [-0.632 to -0.035]

14. Secondary Outcome: Change From Baseline Over Time in the mRESQ-eD Item 'Hoarseness Severity'
Description: The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the severity of their hoarseness over the past 24 hours on a 6-point scale: 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe. Daily scores were averaged each week. A negative change from baseline indicates improvement.
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
units on a scale
  Week 1 | -0.329 (0.074) | -0.292 (0.073) | -0.400 (0.073) | -0.406 (0.074)
  Week 2 | -0.483 (0.090) | -0.416 (0.089) | -0.605 (0.089) | -0.544 (0.091)
  Week 3 | -0.526 (0.095) | -0.574 (0.094) | -0.796 (0.094) | -0.778 (0.096)
  Week 4 | -0.505 (0.102) | -0.631 (0.101) | -0.842 (0.101) | -0.833 (0.103)
  Week 5 | -0.588 (0.107) | -0.684 (0.106) | -0.870 (0.106) | -0.842 (0.108)
  Week 6 | -0.617 (0.110) | -0.677 (0.108) | -0.990 (0.108) | -0.962 (0.110)
  Week 7 | -0.570 (0.111) | -0.626 (0.109) | -0.860 (0.109) | -1.054 (0.111)
  Week 8 | -0.604 (0.108) | -0.683 (0.107) | -0.954 (0.107) | -1.086 (0.109)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.7207, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.037, 95% CI 2-sided [-0.167 to 0.241]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.4946, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.071, 95% CI 2-sided [-0.275 to 0.133]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.4596, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.077, 95% CI 2-sided [-0.283 to 0.129]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.5987, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.067, 95% CI 2-sided [-0.182 to 0.315]
Statistical Analysis 5: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.3348, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.122, 95% CI 2-sided [-0.372 to 0.127]
Statistical Analysis 6: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.6288, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.062, 95% CI 2-sided [-0.313 to 0.190]
Statistical Analysis 7: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.7193, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.048, 95% CI 2-sided [-0.312 to 0.216]
Statistical Analysis 8: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.0452, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.270, 95% CI 2-sided [-0.534 to -0.006]
Statistical Analysis 9: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.0635, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.252, 95% CI 2-sided [-0.519 to 0.014]
Statistical Analysis 10: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.3800, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.126, 95% CI 2-sided [-0.409 to 0.156]
Statistical Analysis 11: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.0200, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.336, 95% CI 2-sided [-0.620 to -0.053]
Statistical Analysis 12: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.0244, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.328, 95% CI 2-sided [-0.614 to -0.043]
Statistical Analysis 13: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.5232, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.096, 95% CI 2-sided [-0.392 to 0.200]
Statistical Analysis 14: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.0623, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.282, 95% CI 2-sided [-0.579 to 0.015]
Statistical Analysis 15: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.0951, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.255, 95% CI 2-sided [-0.554 to 0.045]
Statistical Analysis 16: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.6985, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.060, 95% CI 2-sided [-0.363 to 0.243]
Statistical Analysis 17: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.0163, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.373, 95% CI 2-sided [-0.677 to -0.069]
Statistical Analysis 18: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.0273, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.345, 95% CI 2-sided [-0.652 to -0.039]
Statistical Analysis 19: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.7187, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.056, 95% CI 2-sided [-0.362 to 0.250]
Statistical Analysis 20: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.0640, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.290, 95% CI 2-sided [-0.596 to 0.017]
Statistical Analysis 21: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.0023, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.484, 95% CI 2-sided [-0.793 to -0.175]
Statistical Analysis 22: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.6033, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.079, 95% CI 2-sided [-0.378 to 0.220]
Statistical Analysis 23: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.0222, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.350, 95% CI 2-sided [-0.650 to -0.050]
Statistical Analysis 24: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.0019, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.482, 95% CI 2-sided [-0.785 to -0.180]

15. Secondary Outcome: Change From Baseline Over Time in the mRESQ-eD Item 'Cough Severity'
Description: The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the severity of their cough over the past 24 hours on a 6-point scale: 0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe. Daily scores were averaged each week. A negative change from baseline indicates improvement.
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
units on a scale
  Week 1 | -0.426 (0.078) | -0.283 (0.076) | -0.353 (0.076) | -0.389 (0.078)
  Week 2 | -0.574 (0.095) | -0.501 (0.093) | -0.608 (0.093) | -0.589 (0.095)
  Week 3 | -0.534 (0.092) | -0.614 (0.090) | -0.745 (0.090) | -0.890 (0.092)
  Week 4 | -0.530 (0.099) | -0.657 (0.097) | -0.878 (0.097) | -0.914 (0.099)
  Week 5 | -0.616 (0.106) | -0.692 (0.104) | -0.840 (0.104) | -0.972 (0.107)
  Week 6 | -0.634 (0.107) | -0.671 (0.105) | -0.953 (0.105) | -1.026 (0.107)
  Week 7 | -0.594 (0.112) | -0.688 (0.110) | -0.971 (0.110) | -1.063 (0.112)
  Week 8 | -0.613 (0.107) | -0.706 (0.105) | -0.949 (0.105) | -1.158 (0.107)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.1922, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.143, 95% CI 2-sided [-0.072 to 0.357]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.5091, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.072, 95% CI 2-sided [-0.143 to 0.288]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.7394, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.037, 95% CI 2-sided [-0.181 to 0.254]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.5845, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.073, 95% CI 2-sided [-0.189 to 0.334]
Statistical Analysis 5: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.7959, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.034, 95% CI 2-sided [-0.296 to 0.228]
Statistical Analysis 6: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.9086, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.015, 95% CI 2-sided [-0.280 to 0.249]
Statistical Analysis 7: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.5334, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.080, 95% CI 2-sided [-0.333 to 0.173]
Statistical Analysis 8: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.1020, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.212, 95% CI 2-sided [-0.466 to 0.042]
Statistical Analysis 9: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.0066, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.357, 95% CI 2-sided [-0.613 to -0.100]
Statistical Analysis 10: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.3586, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.127, 95% CI 2-sided [-0.399 to 0.145]
Statistical Analysis 11: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.0128, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.348, 95% CI 2-sided [-0.621 to -0.075]
Statistical Analysis 12: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.0064, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.384, 95% CI 2-sided [-0.660 to -0.109]
Statistical Analysis 13: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.6124, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.076, 95% CI 2-sided [-0.369 to 0.218]
Statistical Analysis 14: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.1365, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.223, 95% CI 2-sided [-0.518 to 0.071]
Statistical Analysis 15: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.0193, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.355, 95% CI 2-sided [-0.652 to -0.058]
Statistical Analysis 16: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.8046, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.037, 95% CI 2-sided [-0.333 to 0.258]
Statistical Analysis 17: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.0350, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.319, 95% CI 2-sided [-0.616 to -0.023]
Statistical Analysis 18: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.0105, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.392, 95% CI 2-sided [-0.691 to -0.093]
Statistical Analysis 19: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.5482, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.094, 95% CI 2-sided [-0.403 to 0.214]
Statistical Analysis 20: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.0170, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.377, 95% CI 2-sided [-0.687 to -0.068]
Statistical Analysis 21: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.0034, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.469, 95% CI 2-sided [-0.781 to -0.157]
Statistical Analysis 22: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.5346, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.093, 95% CI 2-sided [-0.388 to 0.202]
Statistical Analysis 23: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.0262, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.336, 95% CI 2-sided [-0.632 to -0.040]
Statistical Analysis 24: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.0004, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.545, 95% CI 2-sided [-0.843 to -0.246]

16. Secondary Outcome: Change From Baseline Over Time in the mRESQ-eD Item 'Regurgitation Frequency'
Description: The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the frequency of their regurgitation (liquid or food moving upwards towards the throat or mouth) over the past 24 hours on a 5-point scale: 0=Never, 1= Rarely, 2=Sometimes, 3=Often, 4=Very often. Daily scores were averaged each week. A negative change from baseline indicates improvement.
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
units on a scale
  Week 1 | -0.483 (0.067) | -0.385 (0.066) | -0.340 (0.066) | -0.511 (0.068)
  Week 2 | -0.647 (0.082) | -0.637 (0.081) | -0.597 (0.081) | -0.774 (0.083)
  Week 3 | -0.581 (0.084) | -0.784 (0.083) | -0.791 (0.083) | -0.879 (0.085)
  Week 4 | -0.769 (0.089) | -0.855 (0.088) | -0.838 (0.087) | -0.984 (0.089)
  Week 5 | -0.758 (0.087) | -0.869 (0.086) | -0.866 (0.085) | -1.028 (0.087)
  Week 6 | -0.834 (0.090) | -0.936 (0.089) | -0.939 (0.089) | -1.093 (0.090)
  Week 7 | -0.796 (0.090) | -0.899 (0.089) | -0.867 (0.089) | -1.081 (0.091)
  Week 8 | -0.811 (0.092) | -0.951 (0.091) | -1.029 (0.091) | -1.191 (0.093)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.3007, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.098, 95% CI 2-sided [-0.088 to 0.284]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.1295, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.143, 95% CI 2-sided [-0.042 to 0.328]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.7671, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.028, 95% CI 2-sided [-0.216 to 0.159]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.9308, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.010, 95% CI 2-sided [-0.217 to 0.238]
Statistical Analysis 5: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.6595, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.051, 95% CI 2-sided [-0.176 to 0.277]
Statistical Analysis 6: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.2771, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.127, 95% CI 2-sided [-0.356 to 0.102]
Statistical Analysis 7: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.0887, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.203, 95% CI 2-sided [-0.436 to 0.031]
Statistical Analysis 8: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.0758, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.210, 95% CI 2-sided [-0.443 to 0.022]
Statistical Analysis 9: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.0132, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.298, 95% CI 2-sided [-0.534 to -0.063]
Statistical Analysis 10: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.4903, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.086, 95% CI 2-sided [-0.332 to 0.160]
Statistical Analysis 11: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.5824, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.068, 95% CI 2-sided [-0.313 to 0.176]
Statistical Analysis 12: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.0885, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.215, 95% CI 2-sided [-0.463 to 0.033]
Statistical Analysis 13: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.3652, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.111, 95% CI 2-sided [-0.352 to 0.130]
Statistical Analysis 14: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.3739, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.108, 95% CI 2-sided [-0.348 to 0.131]
Statistical Analysis 15: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.0294, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.270, 95% CI 2-sided [-0.512 to -0.027]
Statistical Analysis 16: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.4236, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.102, 95% CI 2-sided [-0.351 to 0.148]
Statistical Analysis 17: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.4071, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.105, 95% CI 2-sided [-0.353 to 0.144]
Statistical Analysis 18: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.0434, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.259, 95% CI 2-sided [-0.510 to -0.008]
Statistical Analysis 19: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.4172, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.103, 95% CI 2-sided [-0.354 to 0.147]
Statistical Analysis 20: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.5759, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.071, 95% CI 2-sided [-0.321 to 0.179]
Statistical Analysis 21: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.0271, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.285, 95% CI 2-sided [-0.538 to -0.033]
Statistical Analysis 22: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.2804, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.140, 95% CI 2-sided [-0.395 to 0.115]
Statistical Analysis 23: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.0913, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.218, 95% CI 2-sided [-0.472 to 0.035]
Statistical Analysis 24: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.0039, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.380, 95% CI 2-sided [-0.637 to -0.123]

17. Secondary Outcome: Change From Baseline Over Time in the mRESQ-eD Item 'Acid or Bitter Taste Frequency'
Description: The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the frequency of an acid or bitter taste in the mouth over the past 24 hours on a 5-point scale: 0=Never, 1= Rarely, 2=Sometimes, 3=Often, 4=Very often. Daily scores were averaged each week. A negative change from baseline indicates improvement.
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
units on a scale
  Week 1 | -0.502 (0.069) | -0.374 (0.068) | -0.401 (0.068) | -0.530 (0.070)
  Week 2 | -0.738 (0.084) | -0.640 (0.082) | -0.676 (0.082) | -0.784 (0.084)
  Week 3 | -0.691 (0.082) | -0.806 (0.081) | -0.842 (0.081) | -0.874 (0.083)
  Week 4 | -0.797 (0.090) | -0.847 (0.088) | -0.893 (0.088) | -0.952 (0.090)
  Week 5 | -0.868 (0.089) | -0.920 (0.087) | -0.929 (0.087) | -1.024 (0.089)
  Week 6 | -0.870 (0.092) | -0.966 (0.091) | -1.009 (0.091) | -1.098 (0.093)
  Week 7 | -0.895 (0.094) | -0.912 (0.092) | -0.947 (0.092) | -1.053 (0.094)
  Week 8 | -0.896 (0.094) | -0.938 (0.093) | -1.072 (0.093) | -1.163 (0.095)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.1902, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.128, 95% CI 2-sided [-0.064 to 0.319]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.3021, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.100, 95% CI 2-sided [-0.091 to 0.292]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.7750, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.028, 95% CI 2-sided [-0.221 to 0.165]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.4022, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.099, 95% CI 2-sided [-0.133 to 0.330]
Statistical Analysis 5: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.5971, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.062, 95% CI 2-sided [-0.169 to 0.293]
Statistical Analysis 6: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.7024, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.045, 95% CI 2-sided [-0.279 to 0.188]
Statistical Analysis 7: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.3173, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.115, 95% CI 2-sided [-0.342 to 0.111]
Statistical Analysis 8: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.1906, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.151, 95% CI 2-sided [-0.378 to 0.076]
Statistical Analysis 9: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.1177, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.183, 95% CI 2-sided [-0.412 to 0.046]
Statistical Analysis 10: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.6936, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.050, 95% CI 2-sided [-0.297 to 0.198]
Statistical Analysis 11: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.4466, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.096, 95% CI 2-sided [-0.343 to 0.152]
Statistical Analysis 12: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.2225, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.155, 95% CI 2-sided [-0.405 to 0.095]
Statistical Analysis 13: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.6764, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.052, 95% CI 2-sided [-0.297 to 0.193]
Statistical Analysis 14: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.6243, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.061, 95% CI 2-sided [-0.306 to 0.184]
Statistical Analysis 15: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.2151, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.156, 95% CI 2-sided [-0.403 to 0.091]
Statistical Analysis 16: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.4611, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.096, 95% CI 2-sided [-0.351 to 0.160]
Statistical Analysis 17: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.2849, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.139, 95% CI 2-sided [-0.394 to 0.116]
Statistical Analysis 18: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.0833, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.228, 95% CI 2-sided [-0.485 to 0.030]
Statistical Analysis 19: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.8955, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.017, 95% CI 2-sided [-0.277 to 0.242]
Statistical Analysis 20: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.6916, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.052, 95% CI 2-sided [-0.312 to 0.207]
Statistical Analysis 21: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.2345, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.159, 95% CI 2-sided [-0.421 to 0.103]
Statistical Analysis 22: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.7466, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.043, 95% CI 2-sided [-0.304 to 0.218]
Statistical Analysis 23: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.1843, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.176, 95% CI 2-sided [-0.437 to 0.084]
Statistical Analysis 24: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.0471, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.267, 95% CI 2-sided [-0.531 to -0.003]

18. Secondary Outcome: Change From Baseline Over Time in the mRESQ-eD Item 'Coughing Frequency'
Description: The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the frequency of their cough over the past 24 hours on a 5-point scale: 0=Never, 1= Rarely, 2=Sometimes, 3=Often, 4=Very often. Daily scores were averaged each week. A negative change from baseline indicates improvement.
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
units on a scale
  Week 1 | -0.374 (0.064) | -0.286 (0.063) | -0.290 (0.063) | -0.352 (0.064)
  Week 2 | -0.572 (0.081) | -0.469 (0.079) | -0.484 (0.079) | -0.571 (0.081)
  Week 3 | -0.477 (0.083) | -0.605 (0.081) | -0.594 (0.081) | -0.729 (0.083)
  Week 4 | -0.497 (0.089) | -0.667 (0.087) | -0.685 (0.087) | -0.793 (0.089)
  Week 5 | -0.506 (0.095) | -0.659 (0.093) | -0.648 (0.093) | -0.812 (0.095)
  Week 6 | -0.594 (0.092) | -0.653 (0.090) | -0.700 (0.090) | -0.872 (0.092)
  Week 7 | -0.561 (0.097) | -0.656 (0.095) | -0.713 (0.095) | -0.872 (0.097)
  Week 8 | -0.554 (0.095) | -0.647 (0.093) | -0.718 (0.093) | -0.988 (0.095)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.3258, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.088, 95% CI 2-sided [-0.088 to 0.265]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.3483, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.084, 95% CI 2-sided [-0.092 to 0.261]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.8055, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.022, 95% CI 2-sided [-0.156 to 0.201]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.3627, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.103, 95% CI 2-sided [-0.119 to 0.326]
Statistical Analysis 5: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.4404, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.087, 95% CI 2-sided [-0.135 to 0.310]
Statistical Analysis 6: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.9939, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.001, 95% CI 2-sided [-0.224 to 0.226]
Statistical Analysis 7: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.2716, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.128, 95% CI 2-sided [-0.356 to 0.100]
Statistical Analysis 8: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.3175, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.116, 95% CI 2-sided [-0.345 to 0.112]
Statistical Analysis 9: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.0325, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.252, 95% CI 2-sided [-0.483 to -0.021]
Statistical Analysis 10: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.1769, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.169, 95% CI 2-sided [-0.415 to 0.077]
Statistical Analysis 11: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.1343, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.188, 95% CI 2-sided [-0.434 to 0.058]
Statistical Analysis 12: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.0203, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.295, 95% CI 2-sided [-0.544 to -0.046]
Statistical Analysis 13: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.2543, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.152, 95% CI 2-sided [-0.415 to 0.110]
Statistical Analysis 14: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.2892, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.142, 95% CI 2-sided [-0.405 to 0.121]
Statistical Analysis 15: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.0243, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.306, 95% CI 2-sided [-0.571 to -0.040]
Statistical Analysis 16: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.6471, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.059, 95% CI 2-sided [-0.312 to 0.194]
Statistical Analysis 17: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.4123, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.106, 95% CI 2-sided [-0.359 to 0.148]
Statistical Analysis 18: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.0338, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.278, 95% CI 2-sided [-0.534 to -0.021]
Statistical Analysis 19: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.4841, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.095, 95% CI 2-sided [-0.362 to 0.172]
Statistical Analysis 20: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.2627, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.152, 95% CI 2-sided [-0.419 to 0.115]
Statistical Analysis 21: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.0241, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.311, 95% CI 2-sided [-0.581 to -0.041]
Statistical Analysis 22: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.4881, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.093, 95% CI 2-sided [-0.355 to 0.170]
Statistical Analysis 23: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.2205, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.164, 95% CI 2-sided [-0.427 to 0.099]
Statistical Analysis 24: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.0015, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.433, 95% CI 2-sided [-0.699 to -0.168]

19. Secondary Outcome: Change From Baseline Over Time in the mRESQ-eD Item 'Burping Frequency'
Description: The mRESQ-eD questionnaire assesses the severity and frequency of the symptoms participants experience due to reflux disease. Participants were asked to rate the frequency of their burping over the past 24 hours on a 5-point scale: 0=Never, 1= Rarely, 2=Sometimes, 3=Often, 4=Very often. Daily scores were averaged each week. A negative change from baseline indicates improvement.
Time Frame: as for outcome 10
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 69 | 71 | 71 | 68
units on a scale
  Week 1 | -0.459 (0.071) | -0.416 (0.070) | -0.309 (0.070) | -0.416 (0.071)
  Week 2 | -0.669 (0.083) | -0.649 (0.082) | -0.556 (0.082) | -0.614 (0.084)
  Week 3 | -0.605 (0.085) | -0.705 (0.084) | -0.734 (0.084) | -0.754 (0.086)
  Week 4 | -0.701 (0.092) | -0.794 (0.091) | -0.797 (0.090) | -0.866 (0.093)
  Week 5 | -0.744 (0.091) | -0.832 (0.090) | -0.813 (0.090) | -0.910 (0.092)
  Week 6 | -0.801 (0.094) | -0.845 (0.093) | -0.845 (0.093) | -0.942 (0.095)
  Week 7 | -0.810 (0.099) | -0.896 (0.098) | -0.803 (0.097) | -0.909 (0.100)
  Week 8 | -0.809 (0.102) | -0.973 (0.101) | -0.920 (0.100) | -1.008 (0.103)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.6653, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.043, 95% CI 2-sided [-0.152 to 0.238]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.1327, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.150, 95% CI 2-sided [-0.046 to 0.345]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 1; Test type: Superiority; p = 0.6697, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.043, 95% CI 2-sided [-0.155 to 0.241]
Statistical Analysis 4: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.8598, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.021, 95% CI 2-sided [-0.210 to 0.251]
Statistical Analysis 5: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.3354, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.113, 95% CI 2-sided [-0.118 to 0.344]
Statistical Analysis 6: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 2; Test type: Superiority; p = 0.6429, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.055, 95% CI 2-sided [-0.179 to 0.289]
Statistical Analysis 7: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.4010, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.101, 95% CI 2-sided [-0.336 to 0.135]
Statistical Analysis 8: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.2821, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.129, 95% CI 2-sided [-0.364 to 0.106]
Statistical Analysis 9: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 3; Test type: Superiority; p = 0.2189, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.149, 95% CI 2-sided [-0.388 to 0.089]
Statistical Analysis 10: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.4717, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.093, 95% CI 2-sided [-0.346 to 0.161]
Statistical Analysis 11: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.4572, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.096, 95% CI 2-sided [-0.349 to 0.158]
Statistical Analysis 12: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 4; Test type: Superiority; p = 0.2064, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.165, 95% CI 2-sided [-0.422 to 0.092]
Statistical Analysis 13: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.4932, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.088, 95% CI 2-sided [-0.339 to 0.164]
Statistical Analysis 14: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.5897, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.069, 95% CI 2-sided [-0.321 to 0.183]
Statistical Analysis 15: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 5; Test type: Superiority; p = 0.2014, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.166, 95% CI 2-sided [-0.421 to 0.089]
Statistical Analysis 16: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.7384, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.044, 95% CI 2-sided [-0.304 to 0.215]
Statistical Analysis 17: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.7423, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.043, 95% CI 2-sided [-0.303 to 0.216]
Statistical Analysis 18: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 6; Test type: Superiority; p = 0.2923, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.141, 95% CI 2-sided [-0.404 to 0.122]
Statistical Analysis 19: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.5388, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.085, 95% CI 2-sided [-0.359 to 0.188]
Statistical Analysis 20: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.9565, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.008, 95% CI 2-sided [-0.266 to 0.281]
Statistical Analysis 21: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 7; Test type: Superiority; p = 0.4848, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.099, 95% CI 2-sided [-0.376 to 0.179]
Statistical Analysis 22: Comparison: Placebo BID vs 500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.2523, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.164, 95% CI 2-sided [-0.445 to 0.117]
Statistical Analysis 23: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.4356, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.112, 95% CI 2-sided [-0.393 to 0.170]
Statistical Analysis 24: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Week 8; Test type: Superiority; p = 0.1706, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.199, 95% CI 2-sided [-0.485 to 0.086]

20. Secondary Outcome: Change From Baseline in the Proportion of Heartburn-Free Days During Week 8
Description: A heartburn free day was a day where DHSS = 0. DHSS was defined as the maximum on a 6-point scale (0=Did Not Have, 1=Very Mild, 2=Mild, 3=Moderate, 4=Moderately Severe, 5=Severe) of the 3 items measuring heartburn ( "Heartburn," "Burning feeling behind breastbone or in the center of the upper stomach," and "Pain behind breastbone or in the center of the upper stomach,") from a particular day.
Time Frame: Week 8
Population: modified Intent-to-Treat Population: all randomized participants who received at least one dose of study treatment with values at treatment week.
Measure: Least Squares Mean (Standard Error); unit: proportion of days
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 61 | 66 | 62 | 62
proportion of days | 0.276 (0.049) | 0.256 (0.047) | 0.310 (0.049) | 0.347 (0.049)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Test type: Superiority; p = 0.7689, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.020, 95% CI 2-sided [-0.155 to 0.115]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Test type: Superiority; p = 0.6287, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.034, 95% CI 2-sided [-0.103 to 0.170]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.3106, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.070, 95% CI 2-sided [-0.066 to 0.207]

21. Secondary Outcome: Change From Baseline in the Proportion of Heartburn-Free Days During Week 4
Description: as for outcome 20
Time Frame: Week 4
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: proportion of days
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
Number analyzed (Participants) | 64 | 70 | 66 | 68
proportion of days | 0.141 (0.037) | 0.142 (0.035) | 0.134 (0.036) | 0.241 (0.036)
Statistical Analysis 1: Comparison: Placebo BID vs 500 mg IW-3718 BID; Test type: Superiority; p = 0.9961, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.000, 95% CI 2-sided [-0.100 to 0.101]
Statistical Analysis 2: Comparison: Placebo BID vs 1000 mg IW-3718 BID; Test type: Superiority; p = 0.8829, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.008, 95% CI 2-sided [-0.109 to 0.094]
Statistical Analysis 3: Comparison: Placebo BID vs 1500 mg IW-3718 BID; Test type: Superiority; p = 0.0527, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.100, 95% CI 2-sided [-0.001 to 0.201]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through Week 8/End-of-treatment (Day 57 + 3 days) plus 7 days.
Description: Treatment-emergent adverse events (TEAEs) are presented. TEAEs are defined as adverse events (AEs) that started after the first dose of study drug or started before the first dose of study drug but increased in severity after the first dose of study drug. Safety population: all participants who were randomized and received at least 1 dose of study drug.
Arm/Group | Placebo BID | 500 mg IW-3718 BID | 1000 mg IW-3718 BID | 1500 mg IW-3718 BID
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/71 | 0/71 | 0/68
Serious Adverse Events (participants affected / at risk) | 2/70 | 1/71 | 1/71 | 2/68
Other Adverse Events (participants affected / at risk) | 16/70 | 17/71 | 19/71 | 12/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID (N=70) | 500 mg IW-3718 BID (N=71) | 1000 mg IW-3718 BID (N=71) | 1500 mg IW-3718 BID (N=68)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Selective abortion (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo BID (N=70) | 500 mg IW-3718 BID (N=71) | 1000 mg IW-3718 BID (N=71) | 1500 mg IW-3718 BID (N=68)
Constipation (Gastrointestinal disorders) | 5 | 6 | 6 | 5
Nausea (Gastrointestinal disorders) | 2 | 3 | 4 | 6
Flatulence (Gastrointestinal disorders) | 3 | 7 | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 2 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 3 | 3
Insomnia (Psychiatric disorders) | 5 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Ironwood. Publication of the results by the Principal Investigator will be subject to mutual agreement between the Investigator and Ironwood.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT02637557/SAP_000.pdf
  • Study Protocol (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT02637557/Prot_001.pdf